CLINICAL TRIAL: NCT03483753
Title: Vasopressin or Norepinephrine in Vasoplegic Shock After Non-cardiac Surgery: a Randomized and Controlled Trial
Brief Title: Vasopressin or Norepinephrine in Vasoplegic Shock After Non-cardiac Surgery
Acronym: VANCSIII
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no funding for the study
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tais Felix Szeles, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 62586316.6.0000.0065
Record Dates: First submitted 2018-02-05; First posted 2018-03-30 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Circulatory Shock; Non-cardiac Surgery
Keywords: Vasopressin; Norepinephrine; Post-operative; Critical Care
MeSH Terms: conditions — Shock; Diabetes Insipidus | interventions — Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vasopressin group (Experimental): Blinded vasopressin
  Interventions: Drug: Vasopressin
- Norepinephrine group (Active Comparator): Blinded norepinephrine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Vasopressin — Blinded Vasopressin will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement.
  Continuous infusion of the drug at doses ranging from 0.01 U / min to 0.06 U / min
  Other Names: Blinded Vasopressin
  Arms: Vasopressin group
Drug: Norepinephrine — Blinded Norepinephrine will be started if there is persistent hypotension, characterized by mean arterial pressure <65 mmHg after fluid replacement. Continuous infusion of the drug at doses ranging from 0.1 mcg / kg / min to 1.0 mcg / kg / min.
  Other Names: Blinded Norepinephrine
  Arms: Norepinephrine group

SUMMARY:
The purpose of the present study is to evaluate the effect of vasopressin compared to norepinephrine on the clinical complications of patients with vasospastic shock after noncardiac surgeries.

DETAILED DESCRIPTION:
The Systemic Inflammatory Response Syndrome (SIRS) is a common complication after non-cardiac surgery, impacting negatively on patient outcome and with high incidence rates. Vasoplegic syndrome is the most serious complication of SIRS and can happen after any type of surgery. The etiology of the vasoplegic syndrome has not yet been fully elucidated, but is known to occur more frequently in patients at high surgical risk, submitted to major surgeries, or in the presence of perioperative complications and patients with comorbidities. In this circumstance, the depletion of vasopressin stocks is described, which may contribute to the refractoriness of the shock and the lack of response to the catecholaminergic drugs. The standard treatment of perioperative vasoplegia has been adequate volume replacement and administration of vasopressors, with norepinephrine being the most commonly used. However, it is known that norepinephrine may have deleterious effects on the body and in 20% of patients with vasospastic shock it is ineffective. Previous studies have suggested benefits of adding vasopressin in refractory situations, especially in septic shock. Recently the VANCS study (Vasopressin or norepinephrine in the vasopregic shock after cardiac surgery: double-blind, controlled and randomized study) demonstrated superiority of vasopressin in the reversion of vasoplegic shock after cardiac surgery, as well as a lower incidence of renal insufficiency, atrial fibrillation and shorter hospitalization time. (Anesthesiology. 2017 Jan;126(1):85-93.)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years;
* Patients undergoing high-risk non-cardiac surgery;
* vasopressor need within 24 hours after surgery, defined as mean arterial pressure (MAP) <65 mmHg after volume resuscitation with at least 1 liter of crystalloid solution (Ringer's lactate) and maintaining a cardiac index> 2.2 ml / min / m²;
* Signature of the informed consent form.

Exclusion Criteria:

* Allergy to vasoactive drugs;
* Previous use of vasopressor;
* Gestation;
* Presence of Raynaud's phenomenon, altered Allen's test, systemic sclerosis or vasospastic diathesis;
* Severe hyponatremia (Na <130 mEq / L);
* Acute mesenteric ischemia;
* Acute coronary syndrome;
* Participation in another study;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence between groups of a composite outcome of all-cause mortality, cardiovascular and renal complications after high-risk non-cardiac surgeries | 30 days
  Cardiovascular complications include: stroke, acute myocardial infarction, cardiogenic shock, nonfatal myocardial injury, and ventricular or supraventricular arrhythmias.
  Renal complications: Acute renal failure with AKIN stage 1 or higher or renal support therapy.

SECONDARY OUTCOMES:
All-cause mortality | 30 days after randomization
  mortality rate of any cause
Acute myocardial infarction | 30 days after randomization
  to compare between groups the incidence of acute myocardial infarction
Cardiogenic shock | 30 days after randomization
  to compare between groups the incidence of cardiogenic shock
Ventricular and / or supraventricular arrhythmia | 30 days
  to compare between groups the incidence of Ventricular and / or supraventricular arrhythmia
Acute respiratory distress syndrome (ARDS) | 30 days
  to compare between groups the incidence of Acute respiratory distress syndrome (ARDS)
Stroke and transient ischemic attack | 30 days
  to compare between groups the incidence of Stroke and transient ischemic attack
Delirium | 30 days
  to compare between groups the incidence of Delirium
Acute renal failure (AKIN 1 or more) | 30 days
  to compare between groups the incidence of Acute renal failure (AKIN 1 or more)
Length of time in the Intensive Care Unit (ICU) and hospital | 30 days
  Length of time in the Intensive Care Unit (ICU) and hospital
Length of mechanical ventilation | 30 days
  Length of mechanical ventilation
Septic shock | 30 days
  to compare between groups the incidence of septic shock
hospital and ICU readmission rate | 30 days
  hospital and ICU readmission rate
Reoperation | 30 days
  number of patients who required reoperation
Incidence of severe adverse events | 30 days
  to compare the incidence of severe adverse outcomes defined as mesenteric ischemia, digital ischemia, hyponatremia (Na<130mEq/L), myocardial infarction or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Juliano P Almeida, MD, PhD, Principal Investigator — University of Sao Paulo; Tais F Szeles, MD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levin MA, Lin HM, Castillo JG, Adams DH, Reich DL, Fischer GW. Early on-cardiopulmonary bypass hypotension and other factors associated with vasoplegic syndrome. Circulation. 2009 Oct 27;120(17):1664-71. doi: 10.1161/CIRCULATIONAHA.108.814533. Epub 2009 Oct 12. PMID 19822810
- [Background] Landry DW, Oliver JA. The pathogenesis of vasodilatory shock. N Engl J Med. 2001 Aug 23;345(8):588-95. doi: 10.1056/NEJMra002709. No abstract available. PMID 11529214
- [Background] Gkisioti S, Mentzelopoulos SD. Vasogenic shock physiology. Open Access Emerg Med. 2011 Jan 6;3:1-6. doi: 10.2147/OAEM.S10388. eCollection 2011. PMID 27147845
- [Background] Teboul JL, Monnet X. Detecting volume responsiveness and unresponsiveness in intensive care unit patients: two different problems, only one solution. Crit Care. 2009;13(4):175. doi: 10.1186/cc7979. Epub 2009 Aug 10. PMID 19678915
- [Background] Brown SM, Lanspa MJ, Jones JP, Kuttler KG, Li Y, Carlson R, Miller RR 3rd, Hirshberg EL, Grissom CK, Morris AH. Survival after shock requiring high-dose vasopressor therapy. Chest. 2013 Mar;143(3):664-671. doi: 10.1378/chest.12-1106. PMID 22911566
- [Background] Morales D, Madigan J, Cullinane S, Chen J, Heath M, Oz M, Oliver JA, Landry DW. Reversal by vasopressin of intractable hypotension in the late phase of hemorrhagic shock. Circulation. 1999 Jul 20;100(3):226-9. doi: 10.1161/01.cir.100.3.226. PMID 10411844
- [Background] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Background] Russell JA. Vasopressin, Norepinephrine, and Vasodilatory Shock after Cardiac Surgery: Another "VASST" Difference? Anesthesiology. 2017 Jan;126(1):9-11. doi: 10.1097/ALN.0000000000001435. No abstract available. PMID 27841820
- [Result] Hajjar LA, Vincent JL, Barbosa Gomes Galas FR, Rhodes A, Landoni G, Osawa EA, Melo RR, Sundin MR, Grande SM, Gaiotto FA, Pomerantzeff PM, Dallan LO, Franco RA, Nakamura RE, Lisboa LA, de Almeida JP, Gerent AM, Souza DH, Gaiane MA, Fukushima JT, Park CL, Zambolim C, Rocha Ferreira GS, Strabelli TM, Fernandes FL, Camara L, Zeferino S, Santos VG, Piccioni MA, Jatene FB, Costa Auler JO Jr, Filho RK. Vasopressin versus Norepinephrine in Patients with Vasoplegic Shock after Cardiac Surgery: The VANCS Randomized Controlled Trial. Anesthesiology. 2017 Jan;126(1):85-93. doi: 10.1097/ALN.0000000000001434. PMID 27841822
- [Result] Takenaka K, Ogawa E, Wada H, Hirata T. Systemic inflammatory response syndrome and surgical stress in thoracic surgery. J Crit Care. 2006 Mar;21(1):48-53; discussion 53-5. doi: 10.1016/j.jcrc.2005.07.001. PMID 16616623
- [Result] Haga Y, Beppu T, Doi K, Nozawa F, Mugita N, Ikei S, Ogawa M. Systemic inflammatory response syndrome and organ dysfunction following gastrointestinal surgery. Crit Care Med. 1997 Dec;25(12):1994-2000. doi: 10.1097/00003246-199712000-00016. PMID 9403749
- [Result] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818